CLINICAL TRIAL: NCT02714179
Title: A Double Blind Randomised Controlled Trial of Preemptive and Preventive Use of Paracetamol for Pain Relief After Cesarean Section
Brief Title: Preemptive and Preventive Use of Paracetamol for Pain Relief After Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Ozlem Ozmete, Medical Doctor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: KA15/80
Record Dates: First submitted 2016-03-14; First posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Cesarean Section; Dehiscence

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Preemptive (Group PE), (Active Comparator): Group I: i.V. paracetamol 1 g (100 ml) was given 30 min before induction of anesthesia.
  Interventions: Drug: Paracetamol was given intravenously in both group at different times
- Group Preventive (Group PV), (Active Comparator): Group II: i.V. paracetamol 1 g (100 ml) was given before the end of surgery.
  Interventions: Drug: Paracetamol was given intravenously in both group at different times

INTERVENTIONS:
Drug: Paracetamol was given intravenously in both group at different times

SUMMARY:
The investigators designed a prospective randomized study to investigate the efficacy of intravenous (IV) preemptive versus preventive paracetamol on postoperative pain scores, patient satisfaction, total morphine consumption and the incidence of morphine-related side effects in patients undergoing cesarean section.

ELIGIBILITY:
Inclusion Criteria:

38 weeks pregnancy, elective cesarean section.

-

Exclusion Criteria:

morbid obesity, cardiac failure, depression.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Visual analog score (VAS) for pain | 24 hours